CLINICAL TRIAL: NCT02414139
Title: A Phase II, Multicenter Study of Oral MET Inhibitor INC280 in Adult Patients With EGFR Wild-type (wt), Advanced Non-small Cell Lung Cancer (NSCLC) (Geometry Mono-1)
Brief Title: Study of Oral cMET Inhibitor INC280 in Patients With EGFR Wild-type (wt), Advanced Non-small Cell Lung Cancer (NSCLC) (Geometry Mono-1)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CINC280A2201; 2014-003850-15 (EudraCT Number)
Record Dates: First submitted 2015-03-31; First posted 2015-04-10 (Estimated); Results first posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-02

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Non Small Cell Lung; Non Small Cell Lung Cancer; Non-small cell lung cancer; NSCLC; INC280; EGFR wild-type (wt); advanced non-small cell lung cancer; advanced/metastatic disease; Non-small cell lung carcinoma (NSCLC); treatment of lung cancer after first metastasis; lung cancer; lung adenocarcinoma; Non small cell lung carcinoma; MET exon 14 deletion; METex14del; MET exon 14 skipping; MET exon 14 mutation; MET mutation; MET amplification; MET inhibitor; MET dysregulation; MET activation; MET signaling; MET pathway; met; cMET; Geometry mono-1; Geometry
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis; Lung Neoplasms; Adenocarcinoma of Lung | interventions — capmatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Cohort 1a: Pre-treated patients with MET GCN ≥ 10 (2/3L) (Experimental): Pre-treated patients with MET GCN ≥ 10 treated with INC280 at 400mg BID as second or third line (2/3L)
  Interventions: Drug: Capmatinib
- Cohort 1b:Pre-treated patients with MET GCN ≥ 6 and < 10 (2/3L) (Experimental): Pre-treated patients with MET GCN ≥ 6 and < 10 treated with INC280 at 400 mg BID as second or third line (2/3L)
  Interventions: Drug: Capmatinib
- Cohort 2: Pre-treated patients with MET GCN ≥ 4 and < 6 (2/3L) (Experimental): Pre-treated patients with MET GCN ≥ 4 and < 6 treated with INC280 at 400mg BID as second or third line (2/3L)
  Interventions: Drug: Capmatinib
- Cohort 3: Pre-treated patients with MET GCN < 4 (2/3L) (Experimental): Pre-treated patients with MET GCN < 4 treated with INC280 at 400mg BID as second or third line (2/3L)
  Interventions: Drug: Capmatinib
- Cohort 4: Pre-treated patients with MET mutation regardless of MET GCN (2/3L) (Experimental): Pre-treated patients with MET mutation regardless of MET GCN treated with INC280 at 400mg BID as second or third line (2/3L)
  Interventions: Drug: Capmatinib
- Cohort 5a: Treatment-naïve patients with MET GCN ≥10 (1L) (Experimental): Treatment-naïve patients with MET GCN ≥10 treated with INC280 at 400mg BID as first-line (1L)
  Interventions: Drug: Capmatinib
- Cohort 5b: Treatment-naïve patients with MET mutation regardless of MET GCN (1L) (Experimental): Treatment-naïve patients with MET mutation regardless of MET GCN treated with INC280 at 400mg BID as first line (1L)
  Interventions: Drug: Capmatinib
- Cohort 6.1 (expansion of Cohort 1a): Pre-treated patients MET GCN ≥ 10 without MET mutation (2L) (Experimental): Pre-treated patients with MET GCN ≥ 10 without MET mutation treated with INC280 at 400 mg BID as second line (2L) (expansion cohort of Cohort 1a)
  Interventions: Drug: Capmatinib
- Cohort 6.2 (expansion of Cohort 4): Pre-treated patients with MET mutation (2L) (Experimental): Pre-treated patients with MET mutation regardless of MET GCN treated with INC280 at 400 mg BID as second line (2L)(expansion of Cohort 4)
  Interventions: Drug: Capmatinib
- Cohort 7 (expansion of Cohort 5b): Treatment-naïve with MET mutation regardless of MET GCN (1L) (Experimental): Treatment-naïve patients with MET mutation regardless of MET GCN treated with INC280 at 400mg BID as first line (1L) (expansion cohort of Cohort 5b)
  Interventions: Drug: Capmatinib

INTERVENTIONS:
Drug: Capmatinib — Capmatinib was administered orally, at a dose of 400 mg on a continuous twice daily dosing schedule.
  Capmatinib was administered to participants in Cohorts 1a, 1b, 2, 3, 4, 5a and 5b in a fasted state. For Cohorts 6.1. 6.2 and 7, capmatinib was administered either with or without food.
  Other Names: INC280

SUMMARY:
Study to evaluate the efficacy and safety of capmatinib as a single-agent treatment for subjects with advanced/metastatic (stage IIIB or IV) non-small cell lung cancer (NSCLC) who had wild-type epidermal growth factor receptor (EGFR wt) (for exon 19 deletions and exon 21 L858R substitution mutations), anaplastic lymphoma kinase (ALK)-negative rearrangement, and mesenchymal epithelial transition (MET) mutations leading to exon 14 deletion (referred to as MET mutation hereafter) and/or MET amplification.

DETAILED DESCRIPTION:
This was a Phase II, multicenter, open-label study. Patients were enrolled in different cohorts based on their MET status (amplification and/or mutation) and prior treatment status: Cohort 1a, Cohort 1b, Cohort 2, Cohort 3, Cohort 4, Cohort 5a, Cohort 5b, Cohort 6, and Cohort 7. MET mutation (by RT-PCR) and/or MET amplification status by gene copy number (GCN, by FISH) was determined by central laboratory.

Patients in Cohorts 1, 2, 3, and 4 had previously failed 1 or 2 prior lines of systemic therapy, while patients enrolled in Cohorts 5 and 7 were treatment-naïve for advanced disease/metastatic disease. Patients enrolled in Cohort 6 had failed 1 prior line of systemic therapy for advanced/ metastatic disease.

Patients with MET mutation were enrolled in Cohort 4 (pre-treated), Cohort 5b (treatment naïve) or Cohort 7 (treatment naïve expansion cohort of Cohort 5b), irrespective of their MET GCN. The enrollment in expansion Cohort 7 started after the completion of enrollment in Cohort 5b.

Patients without MET mutation, were enrolled in Cohorts 1a, 1b, 2, 3 (pre-treated) or 5a (treatment naïve), based on their MET GCN. Patients enrolled in Cohort 6 (expansion cohort of Cohort 1a and Cohort 4) had either MET GCN ≥10 without MET mutation (Cohort 6.1) or MET mutation, irrespective to their MET GCN (Cohort 6.2). The enrollment in Cohort 6 started upon enrollment completion of the respective Cohort 1a or Cohort 4.

All participants in the study received oral capmatinib 400 mg twice daily. A treatment cycle was defined as 21 days. Treatment with capmatinib continued until patient experienced any of the following: disease progression according to RECIST 1.1 as determined by investigator and confirmed by Blinded Independent Review Committee (BIRC), unacceptable toxicity that precluded further treatment, treatment discontinuation at the discretion of the Investigator or patient, lost to follow-up, or death. Treatment with capmatinib was allowed beyond RECIST 1.1-defined disease progression (as determined by investigator and confirmed by BIRC) if, in the judgment of the investigator, there was evidence of clinical benefit and the patient wished to continue on the study treatment. All patients continued to have safety evaluations for 30 days after the last dose of study treatment.

Patients who discontinued treatment with capmatinib for any reason other than disease progression, as determined by the investigator and confirmed by BIRC, death, withdrawal of consent for further assessments, or being lost to follow-up, continued to have tumor assessments (post-treatment efficacy follow-up) until disease progression confirmed by BIRC, death, withdrawal of consent for further assessments, or lost to follow-up.

All patients who discontinued treatment with capmatinib were followed for survival (post-treatment survival follow-up) until death, loss to follow-up, withdrawal of consent to survival follow-up, or the end of the study.

ELIGIBILITY:
Key Inclusion Criteria:

* Subjects with Stage IIIB or IV NSCLC (any histology) at the time of study entry
* Subjects with histologically or cytologically confirmed diagnosis of NSCLC that is:

  1. EGFR wt status (for exon 19 deletions and exon 21 L858R substitution mutations)
  2. and ALK rearrangement-negative
  3. and MET-mutation and/or amplification status (as defined in the protocol).
* For Cohorts 1a, 1b, 2, 3, 4 subjects must have failed one or two prior lines of systemic therapy for advanced disease (stage IIIB or IV NSCLC). For Cohort 6, subjects must have failed one prior line of systemic therapy for advanced disease (stage IIIB or IV NSCLC).
* For Cohorts 5a, 5b, and 7, subjects must not have received any systemic therapy for advanced disease (stage IIIB or IV NSCLC).
* Subjects with at least one measurable lesion as defined by RECIST 1.1. A previously irradiated site lesion may only be counted as a target lesion if there was clear sign of progression since the irradiation.
* Subjects who recovered from all toxicities related to prior anticancer therapies to grade ≤ 1 (Common Terminology Criteria for Adverse Events [CTCAE] v 4.03). Subjects with any grade of alopecia were allowed to enter the study.
* Subjects with adequate organ function
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1

Key Exclusion Criteria:

* Prior treatment with crizotinib, or any other MET or HGF inhibitor
* Characterized EGFR mutations that predict sensitivity to EGFR therapy, including, but not limited to exon 19 deletions and exon 21 mutations.
* Characterized ALK-positive rearrangement.
* Symptomatic central nervous system (CNS) metastases who are neurologically unstable or have required increasing doses of steroids within the 2 weeks prior to study entry to manage CNS symptoms.
* Clinically significant, uncontrolled heart diseases
* Thoracic radiotherapy to lung fields ≤ 4 weeks prior to starting capmatinib or subjects who had not recovered from radiotherapy-related toxicities. For all other anatomic sites (including radiotherapy to thoracic vertebrae and ribs), radiotherapy ≤ 2 weeks prior to starting capmatinib or subjects who had not recovered from radiotherapy-related toxicities.

Palliative radiotherapy for bone lesions ≤ 2 weeks prior to starting capmatinib was allowed.

* Receiving treatment with strong inducers of CYP3A4 and/or any enzyme-inducing anticonvulsant and could not be discontinued ≥ 1 week prior to the start of treatment with capmatinib and for the duration of the study.
* Receiving treatment with unstable or increasing doses of corticosteroids.
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of capmatinib.
* Applicable to Cohorts 1-4 and Cohort 6 only: previous anticancer and investigational agents within 4 weeks or ≤ 5 × half-life of the agent (whichever was longer) before first dose of- capmatinib. If previous treatment was a monoclonal antibody, then the treatment must have been discontinued ≥ 4 weeks before first dose of capmatinib. If previous treatment was an oral targeted agent, then the treatment must have been discontinued ≥ 5 × half-life of the agent before the first dose of capmatinib.
* Pregnant or nursing (lactating) women.
* Women of child-bearing potential, unless they are using highly effective methods of contraception during dosing and for 7 days after stopping treatment
* Sexually active males unless they used a condom during intercourse while taking drug and for 7 days after stopping treatment and should not father a child in this period.
* Presence or history of interstitial lung disease or interstitial pneumonitis, including clinically significant radiation pneumonitis (i.e., affecting activities of daily living or requiring therapeutic intervention).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 373 (Actual)
Dates: Start 2015-06-11 (Actual); Primary Completion 2023-04-12 (Actual); Study Completion 2023-05-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (90):
- United States (13):
  - Pacific Shores Medical Group SC, Long Beach, California
  - University Of California Los Angeles Dept of Onc, Los Angeles, California
  - University of California Irvine Medical Center Chao Family Chao Family Comp Cancer Center, Orange, California
  - H Lee Moffitt Cancer Center and Research Institute ., Tampa, Florida
  - University of Iowa Hospitals and Clinics SC-3, Iowa City, Iowa
  - Massachusetts General Hospital MGH Cancer Center, Boston, Massachusetts
  - VA Ann Arbor Health System VA Ann Arbor Health System, Ann Arbor, Michigan
  - Mayo Clinic Rochester ., Rochester, Minnesota
  - Oregon Health and Science University SC, Portland, Oregon
  - Lehigh Valley Health Network SC, Allentown, Pennsylvania
  - Andrew and Patel Associates, Camp Hill, Pennsylvania
  - Mays Cancer Ctr Uthsa Mdacc SC-5, San Antonio, Texas
  - University of Utah / Huntsman Cancer Institute Oncology, Salt Lake City, Utah
- Argentina (3):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Buenos Aires, Buenos Aires F.D.
  - Novartis Investigative Site, La Rioja
- Novartis Investigative Site, Vienna, Austria
- Novartis Investigative Site, Leuven, Belgium
- France (10):
  - Novartis Investigative Site, Marseille, Bouches Du Rhone
  - Novartis Investigative Site, Dijon, Cote D Or
  - Novartis Investigative Site, Clermont-Ferrand
  - Novartis Investigative Site, La Tronche
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Pierre-Bénite
  - Novartis Investigative Site, Rennes
  - Novartis Investigative Site, Strasbourg
- Germany (14):
  - Novartis Investigative Site, Heidelberg, Baden-Wurttemberg
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Göttingen
  - Novartis Investigative Site, Halle
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Homburg
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Nuremberg
  - Novartis Investigative Site, Ravensburg
  - Novartis Investigative Site, Tübingen
  - Novartis Investigative Site, Ulm
- Israel (2):
  - Novartis Investigative Site, Ramat Gan
  - Novartis Investigative Site, Tel Aviv
- Italy (12):
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Brescia, BS
  - Novartis Investigative Site, Catania, CT
  - Novartis Investigative Site, Catanzaro, CZ
  - Novartis Investigative Site, Meldola, FC
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Monza, MB
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Modena, MO
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Verona, VR
  - Novartis Investigative Site, Napoli
- Japan (9):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Akashi, Hyōgo
  - Novartis Investigative Site, Sendai, Miyagi
  - Novartis Investigative Site, Okayama, Okayama-ken
  - Novartis Investigative Site, Ōsaka-sayama, Osaka
  - Novartis Investigative Site, Chuo Ku, Tokyo
  - Novartis Investigative Site, Koto Ku, Tokyo
  - Novartis Investigative Site, Ube, Yamaguchi
- Novartis Investigative Site, El Achrafiyé, Lebanon
- Novartis Investigative Site, Mexico City, Mexico City, Mexico
- Netherlands (4):
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Groningen
  - Novartis Investigative Site, Maastricht
  - Novartis Investigative Site, Rotterdam
- Novartis Investigative Site, Oslo, Norway
- Russia (3):
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Tambov
- Novartis Investigative Site, Singapore, Singapore
- South Korea (3):
  - Novartis Investigative Site, Bundang Gu, Gyeonggi-do
  - Novartis Investigative Site, Gyeonggi-do, Korea
  - Novartis Investigative Site, Seoul
- Spain (5):
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, A Coruña, Galicia
  - Novartis Investigative Site, Oviedo, Principality of Asturias
  - Novartis Investigative Site, Madrid
- Novartis Investigative Site, Stockholm, Sweden
- Taiwan (3):
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Taipei
  - Novartis Investigative Site, Taoyuan District
- United Kingdom (2):
  - Novartis Investigative Site, Birmingham
  - Novartis Investigative Site, London

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Wolf J, Hochmair M, Han JY, Reguart N, Souquet PJ, Smit EF, Orlov SV, Vansteenkiste J, Nishio M, de Jonge M, Akerley W, Garon EB, Groen HJM, Tan DSW, Seto T, Frampton GM, Robeva A, Carbini M, Le Mouhaer S, Yovine A, Boran A, Bossen C, Yang Y, Ji L, Fairchild L, Heist RS. Capmatinib in MET exon 14-mutated non-small-cell lung cancer: final results from the open-label, phase 2 GEOMETRY mono-1 trial. Lancet Oncol. 2024 Oct;25(10):1357-1370. doi: 10.1016/S1470-2045(24)00441-8. PMID 39362249
- [Derived] Wolf J, Garon EB, Groen HJM, Tan DSW, Gilloteau I, Le Mouhaer S, Hampe M, Cai C, Chassot-Agostinho A, Reynolds M, Sherif B, Heist RS. Patient-reported outcomes in capmatinib-treated patients with METex14-mutated advanced NSCLC: Results from the GEOMETRY mono-1 study. Eur J Cancer. 2023 Apr;183:98-108. doi: 10.1016/j.ejca.2022.10.030. Epub 2022 Dec 10. PMID 36822130
- [Derived] Wolf J, Seto T, Han JY, Reguart N, Garon EB, Groen HJM, Tan DSW, Hida T, de Jonge M, Orlov SV, Smit EF, Souquet PJ, Vansteenkiste J, Hochmair M, Felip E, Nishio M, Thomas M, Ohashi K, Toyozawa R, Overbeck TR, de Marinis F, Kim TM, Laack E, Robeva A, Le Mouhaer S, Waldron-Lynch M, Sankaran B, Balbin OA, Cui X, Giovannini M, Akimov M, Heist RS; GEOMETRY mono-1 Investigators. Capmatinib in MET Exon 14-Mutated or MET-Amplified Non-Small-Cell Lung Cancer. N Engl J Med. 2020 Sep 3;383(10):944-957. doi: 10.1056/NEJMoa2002787. PMID 32877583
- See also: For interim results on this study, please click the link below to the NovartisClinicalTrial.com website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17663

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in 95 centers across 20 countries
Pre-assignment Details: Screening assessments were conducted up to 28 days prior to the start of study treatment
Groups:
- Cohort 1b: Pre-treated Patients With MET GCN ≥ 6 and < 10 (2/3L): Pre-treated patients with MET GCN ≥ 6 and < 10 treated with INC280 at 400 mg BID as second or third line (2/3L)
Period: Treatment Period
Arm/Group | Cohort 1a: Pre-treated Patients With MET GCN ≥ 10 (2/3L) | Cohort 1b: Pre-treated Patients With MET GCN ≥ 6 and < 10 (2/3L) | Cohort 2: Pre-treated Patients With MET GCN ≥ 4 and < 6 (2/3L) | Cohort 3: Pre-treated Patients With MET GCN < 4 (2/3L) | Cohort 4: Pre-treated Patients With MET Mutation Regardless of MET GCN (2/3L) | Cohort 5a: Treatment-naïve Patients With MET GCN ≥10 (1L) | Cohort 5b: Treatment-naïve Patients With MET Mutation Regardless of MET GCN (1L) | Cohort 6.1 (Expansion of Cohort 1a): Pre-treated Patients MET GCN ≥ 10 Without MET Mutation (2L) | Cohort 6.2 (Expansion of Cohort 4): Pre-treated Patients With MET Mutation (2L) | Cohort 7 (Expansion of Cohort 5b): Treatment-naïve With MET Mutation Regardless of MET GCN (1L)
Started | 69 | 42 | 54 | 30 | 69 | 15 | 28 | 3 | 31 | 32
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 69 | 42 | 54 | 30 | 69 | 15 | 28 | 3 | 31 | 32
Not completed — Adverse Event | 11 | 6 | 8 | 5 | 14 | 3 | 6 | 1 | 6 | 8
Not completed — Death | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Physician Decision | 5 | 4 | 6 | 1 | 4 | 0 | 2 | 0 | 1 | 4
Not completed — Progressive disease | 48 | 31 | 37 | 21 | 43 | 12 | 16 | 2 | 20 | 14
Not completed — Protocol deviation | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Subject/Guardian decision | 5 | 1 | 1 | 2 | 5 | 0 | 2 | 0 | 1 | 1
Not completed — Study terminated (as per protocol) by Sponsor | 0 | 0 | 0 | 0 | 3 | 0 | 2 | 0 | 3 | 4
Period: Post-treatment Efficacy Follow-up
Arm/Group | Cohort 1a: Pre-treated Patients With MET GCN ≥ 10 (2/3L) | Cohort 1b: Pre-treated Patients With MET GCN ≥ 6 and < 10 (2/3L) | Cohort 2: Pre-treated Patients With MET GCN ≥ 4 and < 6 (2/3L) | Cohort 3: Pre-treated Patients With MET GCN < 4 (2/3L) | Cohort 4: Pre-treated Patients With MET Mutation Regardless of MET GCN (2/3L) | Cohort 5a: Treatment-naïve Patients With MET GCN ≥10 (1L) | Cohort 5b: Treatment-naïve Patients With MET Mutation Regardless of MET GCN (1L) | Cohort 6.1 (Expansion of Cohort 1a): Pre-treated Patients MET GCN ≥ 10 Without MET Mutation (2L) | Cohort 6.2 (Expansion of Cohort 4): Pre-treated Patients With MET Mutation (2L) | Cohort 7 (Expansion of Cohort 5b): Treatment-naïve With MET Mutation Regardless of MET GCN (1L)
Started | 16 | 11 | 16 | 8 | 23 | 5 | 6 | 1 | 3 | 8
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 16 | 11 | 16 | 8 | 23 | 5 | 6 | 1 | 3 | 8
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 4 | 2 | 4 | 2 | 4 | 0 | 1 | 0 | 0 | 1
Not completed — Progressive disease | 6 | 5 | 9 | 5 | 15 | 4 | 5 | 1 | 3 | 3
Not completed — Study terminated by sponsor | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Subject/guardian decision | 4 | 2 | 3 | 1 | 1 | 1 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1a: Pre-treated Patients With MET GCN ≥ 10 (2/3L) | Cohort 1b: Pre-treated Patients With MET GCN ≥ 6 and < 10 (2/3L) | Cohort 2: Pre-treated Patients With MET GCN ≥ 4 and < 6 (2/3L) | Cohort 3: Pre-treated Patients With MET GCN < 4 (2/3L) | Cohort 4: Pre-treated Patients With MET Mutation Regardless of MET GCN (2/3L) | Cohort 5a: Treatment-naïve Patients With MET GCN ≥10 (1L) | Cohort 5b: Treatment-naïve Patients With MET Mutation Regardless of MET GCN (1L) | Cohort 6.1 (Expansion of Cohort 1a): Pre-treated Patients MET GCN ≥ 10 Without MET Mutation (2L) | Cohort 6.2 (Expansion of Cohort 4): Pre-treated Patients With MET Mutation (2L) | Cohort 7 (Expansion of Cohort 5b): Treatment-naïve With MET Mutation Regardless of MET GCN (1L) | Total
Number analyzed (Participants) | 69 | 42 | 54 | 30 | 69 | 15 | 28 | 3 | 31 | 32 | 373
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.9 (9.56) | 59.5 (9.11) | 61.7 (10.00) | 61.7 (9.23) | 71.0 (8.32) | 68.2 (10.36) | 72.4 (7.02) | 60.7 (10.69) | 69.0 (6.29) | 73.3 (8.35) | 65.7 (10.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 21 | 15 | 11 | 40 | 4 | 18 | 1 | 16 | 23 | 164
  Male | 54 | 21 | 39 | 19 | 29 | 11 | 10 | 2 | 15 | 9 | 209
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 17 | 4 | 14 | 11 | 19 | 6 | 4 | 1 | 5 | 3 | 84
  Black | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3
  Caucasian | 51 | 38 | 40 | 19 | 49 | 9 | 24 | 1 | 24 | 26 | 281
  Native American | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2
  Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) by Blinded Independent Review Committee (BIRC) Assessment
Description: Percentage of participants with a best overall response defined as confirmed complete response (CR) or partial response (PR) by BIRC assessment per RECIST 1.1.
  CR: Disappearance of all non-nodal target and non-target lesions. In addition, any pathological lymph nodes assigned as target and non-target lesions must have a reduction in short axis to < 10 mm PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: Up to approximately 5 years
Population: Full Analysis Set (FAS)-including all subjects who received at least one dose of capmatinib
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Cohort 4 + Cohort 6.2: All Pre-treated Patients With MET Mutation Regardless of MET GCN (2/3L): All pre-treated patients with MET mutation regardless of MET GCN treated with INC280 at 400mg BID as second or third line (2/3L). (Participants from Cohort 4 and Cohort 6.2)
- Cohort 5b + Cohort 7: All Treatment-naive With MET Mutation Regardless of MET GCN (1L): All treatment naive patients with MET mutation regardless of MET GCN treated with INC280 at 400 mg BID as first line (1L) (Participants from Cohort 5b and Cohort 7)
Arm/Group | Cohort 1a: Pre-treated Patients With MET GCN ≥ 10 (2/3L) | Cohort 1b: Pre-treated Patients With MET GCN ≥ 6 and < 10 (2/3L) | Cohort 2: Pre-treated Patients With MET GCN ≥ 4 and < 6 (2/3L) | Cohort 3: Pre-treated Patients With MET GCN < 4 (2/3L) | Cohort 4: Pre-treated Patients With MET Mutation Regardless of MET GCN (2/3L) | Cohort 5a: Treatment-naïve Patients With MET GCN ≥10 (1L) | Cohort 5b: Treatment-naïve Patients With MET Mutation Regardless of MET GCN (1L) | Cohort 6.1 (Expansion of Cohort 1a): Pre-treated Patients MET GCN ≥ 10 Without MET Mutation (2L) | Cohort 6.2 (Expansion of Cohort 4): Pre-treated Patients With MET Mutation (2L) | Cohort 7 (Expansion of Cohort 5b): Treatment-naïve With MET Mutation Regardless of MET GCN (1L) | Cohort 4 + Cohort 6.2: All Pre-treated Patients With MET Mutation Regardless of MET GCN (2/3L) | Cohort 5b + Cohort 7: All Treatment-naive With MET Mutation Regardless of MET GCN (1L)
Number analyzed (Participants) | 69 | 42 | 54 | 30 | 69 | 15 | 28 | 3 | 31 | 32 | 100 | 60
Percentage of Participants | 29.0 [18.7 to 41.2] | 11.9 [4.0 to 25.6] | 9.3 [3.1 to 20.3] | 6.7 [0.8 to 22.1] | 40.6 [28.9 to 53.1] | 40.0 [16.3 to 67.7] | 67.9 [47.6 to 84.1] | 0.0 [0.0 to 70.8] | 51.6 [33.1 to 69.8] | 68.8 [50.0 to 83.9] | 44.0 [34.1 to 54.3] | 68.3 [55.0 to 79.7]

2. Secondary Outcome: Duration of Response (DOR) by BIRC Assessment
Description: Time from the date of the first documented CR or PR by BIRC per RECIST 1.1 to the first documented progression or date of death due to any cause for patients with confirmed PR or CR. The Kaplan-Meier method was used to estimate DOR, and the median DOR, along with 95% confidence intervals was reported. If a subject did not have an event, DOR was censored at the date of last adequate tumor assessment.
  CR: Disappearance of all non-nodal target and non-target lesions. In addition, any pathological lymph nodes assigned as target and non-target lesions must have a reduction in short axis to < 10 mm.
  PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: Up to approximately 5 years
Population: Participants with confirmed CR or PR by BIRC in FAS
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1a: Pre-treated Patients With MET GCN ≥ 10 (2/3L) | Cohort 1b: Pre-treated Patients With MET GCN ≥ 6 and < 10 (2/3L) | Cohort 2: Pre-treated Patients With MET GCN ≥ 4 and < 6 (2/3L) | Cohort 3: Pre-treated Patients With MET GCN < 4 (2/3L) | Cohort 4: Pre-treated Patients With MET Mutation Regardless of MET GCN (2/3L) | Cohort 5a: Treatment-naïve Patients With MET GCN ≥10 (1L) | Cohort 5b: Treatment-naïve Patients With MET Mutation Regardless of MET GCN (1L) | Cohort 6.1 (Expansion of Cohort 1a): Pre-treated Patients MET GCN ≥ 10 Without MET Mutation (2L) | Cohort 6.2 (Expansion of Cohort 4): Pre-treated Patients With MET Mutation (2L) | Cohort 7 (Expansion of Cohort 5b): Treatment-naïve With MET Mutation Regardless of MET GCN (1L) | Cohort 4 + Cohort 6.2: All Pre-treated Patients With MET Mutation Regardless of MET GCN (2/3L) | Cohort 5b + Cohort 7: All Treatment-naive With MET Mutation Regardless of MET GCN (1L)
Number analyzed (Participants) | 20 | 5 | 5 | 2 | 28 | 6 | 19 | 0 | 16 | 22 | 44 | 41
Months | 8.31 [4.17 to 15.44] | 24.94 [2.69 to 24.94] | 9.66 [4.17 to NA] — NA: not estimable due to the insufficient number of participants with events | 4.19 [4.17 to 4.21] | 9.72 [5.55 to 12.98] | 7.54 [2.56 to 14.26] | 12.58 [5.55 to 38.67] |  | 9.05 [4.17 to 27.60] | 16.59 [8.34 to NA] — NA: not estimable due to the insufficient number of participants with events | 9.72 [5.62 to 12.98] | 16.59 [8.41 to 22.11]

3. Secondary Outcome: ORR by Investigator Assessment
Description: Percentage of patients with a best overall response defined as confirmed CR or PR per RECIST 1.1 by investigator assessment.
  CR: Disappearance of all non-nodal target and non-target lesions. In addition, any pathological lymph nodes assigned as target and non-target lesions must have a reduction in short axis to < 10 mm.
  PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: Up to approximately 5 years
Population: FAS, including all subjects who received at least one dose of capmatinib.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1a: Pre-treated Patients With MET GCN ≥ 10 (2/3L) | Cohort 1b: Pre-treated Patients With MET GCN ≥ 6 and < 10 (2/3L) | Cohort 2: Pre-treated Patients With MET GCN ≥ 4 and < 6 (2/3L) | Cohort 3: Pre-treated Patients With MET GCN < 4 (2/3L) | Cohort 4: Pre-treated Patients With MET Mutation Regardless of MET GCN (2/3L) | Cohort 5a: Treatment-naïve Patients With MET GCN ≥10 (1L) | Cohort 5b: Treatment-naïve Patients With MET Mutation Regardless of MET GCN (1L) | Cohort 6.1 (Expansion of Cohort 1a): Pre-treated Patients MET GCN ≥ 10 Without MET Mutation (2L) | Cohort 6.2 (Expansion of Cohort 4): Pre-treated Patients With MET Mutation (2L) | Cohort 7 (Expansion of Cohort 5b): Treatment-naïve With MET Mutation Regardless of MET GCN (1L) | Cohort 4 + Cohort 6.2: All Pre-treated Patients With MET Mutation Regardless of MET GCN (2/3L) | Cohort 5b + Cohort 7: All Treatment-naive With MET Mutation Regardless of MET GCN (1L)
Number analyzed (Participants) | 69 | 42 | 54 | 30 | 69 | 15 | 28 | 3 | 31 | 32 | 100 | 60
Percentage of participants | 27.5 [17.5 to 39.6] | 7.1 [1.5 to 19.5] | 9.3 [3.1 to 20.3] | 3.3 [0.1 to 17.2] | 43.5 [31.6 to 56.0] | 40.0 [16.3 to 67.7] | 60.7 [40.6 to 78.5] | 0.0 [0.0 to 70.8] | 45.2 [27.3 to 64.0] | 56.3 [37.7 to 73.6] | 44.0 [34.1 to 54.3] | 58.3 [44.9 to 70.9]

4. Secondary Outcome: DOR by Investigator Assessment
Description: Time from the date of the first documented CR or PR per RECIST 1.1 by investigator assessment to the first documented progression or death due to any cause for patients with confirmed PR or CR. The Kaplan-Meier method was used to estimate DOR, and the median DOR, along with 95% confidence intervals was reported. If a subject did not have an event, DOR was censored at the date of last adequate tumor assessment.
  CR: Disappearance of all non-nodal target and non-target lesions. In addition, any pathological lymph nodes assigned as target and non-target lesions must have a reduction in short axis to < 10 mm.
  PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: Up to approximately 5 years
Population: Participants with confirmed CR or PR by investigator assessment in FAS.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1a: Pre-treated Patients With MET GCN ≥ 10 (2/3L) | Cohort 1b: Pre-treated Patients With MET GCN ≥ 6 and < 10 (2/3L) | Cohort 2: Pre-treated Patients With MET GCN ≥ 4 and < 6 (2/3L) | Cohort 3: Pre-treated Patients With MET GCN < 4 (2/3L) | Cohort 4: Pre-treated Patients With MET Mutation Regardless of MET GCN (2/3L) | Cohort 5a: Treatment-naïve Patients With MET GCN ≥10 (1L) | Cohort 5b: Treatment-naïve Patients With MET Mutation Regardless of MET GCN (1L) | Cohort 6.1 (Expansion of Cohort 1a): Pre-treated Patients MET GCN ≥ 10 Without MET Mutation (2L) | Cohort 6.2 (Expansion of Cohort 4): Pre-treated Patients With MET Mutation (2L) | Cohort 7 (Expansion of Cohort 5b): Treatment-naïve With MET Mutation Regardless of MET GCN (1L) | Cohort 4 + Cohort 6.2: All Pre-treated Patients With MET Mutation Regardless of MET GCN (2/3L) | Cohort 5b + Cohort 7: All Treatment-naive With MET Mutation Regardless of MET GCN (1L)
Number analyzed (Participants) | 19 | 3 | 5 | 1 | 30 | 6 | 17 | 0 | 14 | 18 | 44 | 35
Months | 6.80 [4.21 to 20.73] | 6.93 [5.75 to 8.34] | 19.48 [2.83 to NA] — NA: not estimable due to the insufficient number of participants with events | 6.93 [NA to NA] — NA: not estimable due to the insufficient number of participants with events | 8.31 [4.34 to 12.06] | 9.66 [4.01 to 17.08] | 13.83 [4.27 to 25.33] |  | 14.57 [4.17 to 27.60] | 15.21 [6.77 to 31.77] | 8.38 [5.55 to 13.80] | 13.96 [9.33 to 22.18]

5. Secondary Outcome: Time to Response (TTR) by BIRC Assessment
Description: Time between date of start of treatment until first documented response (confirmed CR or PR) per RECIST 1.1 by BIRC assessment.
  CR: Disappearance of all non-nodal target and non-target lesions. In addition, any pathological lymph nodes assigned as target and non-target lesions must have a reduction in short axis to < 10 mm.
  PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: Up to approximately 5 years
Population: Participants with confirmed CR or PR by BIRC in FAS
Measure: Median (Full Range); unit: Months
Arm/Group | Cohort 1a: Pre-treated Patients With MET GCN ≥ 10 (2/3L) | Cohort 1b: Pre-treated Patients With MET GCN ≥ 6 and < 10 (2/3L) | Cohort 2: Pre-treated Patients With MET GCN ≥ 4 and < 6 (2/3L) | Cohort 3: Pre-treated Patients With MET GCN < 4 (2/3L) | Cohort 4: Pre-treated Patients With MET Mutation Regardless of MET GCN (2/3L) | Cohort 5a: Treatment-naïve Patients With MET GCN ≥10 (1L) | Cohort 5b: Treatment-naïve Patients With MET Mutation Regardless of MET GCN (1L) | Cohort 6.1 (Expansion of Cohort 1a): Pre-treated Patients MET GCN ≥ 10 Without MET Mutation (2L) | Cohort 6.2 (Expansion of Cohort 4): Pre-treated Patients With MET Mutation (2L) | Cohort 7 (Expansion of Cohort 5b): Treatment-naïve With MET Mutation Regardless of MET GCN (1L) | Cohort 4 + Cohort 6.2: All Pre-treated Patients With MET Mutation Regardless of MET GCN (2/3L) | Cohort 5b + Cohort 7: All Treatment-naive With MET Mutation Regardless of MET GCN (1L)
Number analyzed (Participants) | 20 | 5 | 5 | 2 | 28 | 6 | 19 | 0 | 16 | 22 | 44 | 41
Months | 1.4 [0.5 to 6.8] | 2.8 [1.4 to 16.6] | 1.4 [1.2 to 6.2] | 3.4 [1.3 to 5.5] | 1.4 [1.2 to 5.6] | 1.4 [1.2 to 2.9] | 1.4 [1.3 to 6.9] |  | 1.4 [1.1 to 9.8] | 1.4 [1.2 to 7.2] | 1.4 [1.1 to 9.8] | 1.4 [1.2 to 7.2]

6. Secondary Outcome: TTR by Investigator Assessment
Description: Time between date of start of treatment until first documented response (confirmed CR or PR) per RECIST 1.1 by investigator assessment.
  CR: Disappearance of all non-nodal target and non-target lesions. In addition, any pathological lymph nodes assigned as target and non-target lesions must have a reduction in short axis to < 10 mm.
  PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: Up to approximately 5 years
Population: Participants with confirmed CR or PR by investigator assessment in FAS
Measure: Median (Full Range); unit: Months
Arm/Group | Cohort 1a: Pre-treated Patients With MET GCN ≥ 10 (2/3L) | Cohort 1b: Pre-treated Patients With MET GCN ≥ 6 and < 10 (2/3L) | Cohort 2: Pre-treated Patients With MET GCN ≥ 4 and < 6 (2/3L) | Cohort 3: Pre-treated Patients With MET GCN < 4 (2/3L) | Cohort 4: Pre-treated Patients With MET Mutation Regardless of MET GCN (2/3L) | Cohort 5a: Treatment-naïve Patients With MET GCN ≥10 (1L) | Cohort 5b: Treatment-naïve Patients With MET Mutation Regardless of MET GCN (1L) | Cohort 6.1 (Expansion of Cohort 1a): Pre-treated Patients MET GCN ≥ 10 Without MET Mutation (2L) | Cohort 6.2 (Expansion of Cohort 4): Pre-treated Patients With MET Mutation (2L) | Cohort 7 (Expansion of Cohort 5b): Treatment-naïve With MET Mutation Regardless of MET GCN (1L) | Cohort 4 + Cohort 6.2: All Pre-treated Patients With MET Mutation Regardless of MET GCN (2/3L) | Cohort 5b + Cohort 7: All Treatment-naive With MET Mutation Regardless of MET GCN (1L)
Number analyzed (Participants) | 19 | 3 | 5 | 1 | 30 | 6 | 17 | 0 | 14 | 18 | 44 | 35
Months | 1.4 [1.2 to 5.4] | 1.4 [1.3 to 1.4] | 1.3 [1.2 to 1.7] | 1.3 [1.3 to 1.3] | 1.4 [1.2 to 11.1] | 1.4 [1.3 to 2.5] | 1.4 [1.2 to 4.0] |  | 1.4 [1.1 to 12.3] | 1.4 [1.2 to 5.6] | 1.4 [1.1 to 12.3] | 1.4 [1.2 to 5.6]

7. Secondary Outcome: Disease Control Rate (DCR)
Description: Percentage of participants with a best overall response of confirmed CR, PR or stable disease (SD) per RECIST 1.1 by BIRC and investigator assessment.
  CR: Disappearance of all non-nodal target and non-target lesions. In addition, any pathological lymph nodes assigned as target and non-target lesions must have a reduction in short axis to < 10 mm.
  PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
  SD: Neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions which would qualify for progressive disease.
Time Frame: Up to approximately 5 years
Population: FAS, including all subjects who received at least one dose of capmatinib.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1a: Pre-treated Patients With MET GCN ≥ 10 (2/3L) | Cohort 1b: Pre-treated Patients With MET GCN ≥ 6 and < 10 (2/3L) | Cohort 2: Pre-treated Patients With MET GCN ≥ 4 and < 6 (2/3L) | Cohort 3: Pre-treated Patients With MET GCN < 4 (2/3L) | Cohort 4: Pre-treated Patients With MET Mutation Regardless of MET GCN (2/3L) | Cohort 5a: Treatment-naïve Patients With MET GCN ≥10 (1L) | Cohort 5b: Treatment-naïve Patients With MET Mutation Regardless of MET GCN (1L) | Cohort 6.1 (Expansion of Cohort 1a): Pre-treated Patients MET GCN ≥ 10 Without MET Mutation (2L) | Cohort 6.2 (Expansion of Cohort 4): Pre-treated Patients With MET Mutation (2L) | Cohort 7 (Expansion of Cohort 5b): Treatment-naïve With MET Mutation Regardless of MET GCN (1L) | Cohort 4 + Cohort 6.2: All Pre-treated Patients With MET Mutation Regardless of MET GCN (2/3L) | Cohort 5b + Cohort 7: All Treatment-naive With MET Mutation Regardless of MET GCN (1L)
Number analyzed (Participants) | 69 | 42 | 54 | 30 | 69 | 15 | 28 | 3 | 31 | 32 | 100 | 60
Percentage of participants
  By BIRC assessment | 71.0 [58.8 to 81.3] | 54.8 [38.7 to 70.2] | 46.3 [32.6 to 60.4] | 53.3 [34.3 to 71.7] | 78.3 [66.7 to 87.3] | 66.7 [38.4 to 88.2] | 96.4 [81.7 to 99.9] | 100.0 [29.2 to 100.0] | 90.3 [74.2 to 98.0] | 100.0 [89.1 to 100.0] | 82.0 [73.1 to 89.0] | 98.3 [91.1 to 100.0]
  By investigator assessment | 60.9 [48.4 to 72.4] | 45.2 [29.8 to 61.3] | 44.4 [30.9 to 58.6] | 46.7 [28.3 to 65.7] | 76.8 [65.1 to 86.1] | 73.3 [44.9 to 92.2] | 96.4 [81.7 to 99.9] | 100.0 [29.2 to 100.0] | 90.3 [74.2 to 98.0] | 96.9 [83.8 to 99.9] | 81.0 [71.9 to 88.2] | 96.7 [88.5 to 99.6]

8. Secondary Outcome: Progression-Free Survival
Description: Time from start of treatment to the date of the first documented progression or death due to any cause per RECIST 1.1 by BIRC and investigator assessment. Clinical deterioration was not considered as a qualifying event for progression. PFS was censored at the last adequate tumor assessment if one of the following occurred: absence of event or the event occurred after two or more missing tumor assessments.
  The Kaplan-Meier method was used to estimate PFS, and the median PFS, along with 95% confidence intervals, was reported.
  Progressive disease: For target lesions, at least a 20% increase in the sum of diameter of all measured target lesions, taking as reference the smallest sum of diameter of all target lesions recorded at or after baseline. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm^2. For non-target lesions, unequivocal progression of existing non-target lesions
Time Frame: Up to approximately 5 years
Population: FAS, including all subjects who received at least one dose of capmatinib.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1a: Pre-treated Patients With MET GCN ≥ 10 (2/3L) | Cohort 1b: Pre-treated Patients With MET GCN ≥ 6 and < 10 (2/3L) | Cohort 2: Pre-treated Patients With MET GCN ≥ 4 and < 6 (2/3L) | Cohort 3: Pre-treated Patients With MET GCN < 4 (2/3L) | Cohort 4: Pre-treated Patients With MET Mutation Regardless of MET GCN (2/3L) | Cohort 5a: Treatment-naïve Patients With MET GCN ≥10 (1L) | Cohort 5b: Treatment-naïve Patients With MET Mutation Regardless of MET GCN (1L) | Cohort 6.1 (Expansion of Cohort 1a): Pre-treated Patients MET GCN ≥ 10 Without MET Mutation (2L) | Cohort 6.2 (Expansion of Cohort 4): Pre-treated Patients With MET Mutation (2L) | Cohort 7 (Expansion of Cohort 5b): Treatment-naïve With MET Mutation Regardless of MET GCN (1L) | Cohort 4 + Cohort 6.2: All Pre-treated Patients With MET Mutation Regardless of MET GCN (2/3L) | Cohort 5b + Cohort 7: All Treatment-naive With MET Mutation Regardless of MET GCN (1L)
Number analyzed (Participants) | 69 | 42 | 54 | 30 | 69 | 15 | 28 | 3 | 31 | 32 | 100 | 60
Months
  By BIRC assessment | 4.07 [2.86 to 4.83] | 2.66 [1.41 to 3.09] | 2.66 [1.41 to 4.14] | 3.55 [2.20 to 4.21] | 5.42 [4.17 to 6.97] | 4.17 [1.45 to 6.87] | 12.42 [8.21 to 23.39] | 2.79 [2.07 to 4.24] | 6.93 [4.17 to 13.34] | 12.45 [6.87 to 22.05] | 5.49 [4.17 to 8.11] | 12.45 [8.31 to 17.97]
  By investigator assessment | 4.14 [2.79 to 5.52] | 2.40 [1.45 to 2.83] | 2.60 [1.48 to 3.09] | 2.73 [1.45 to 3.78] | 4.80 [4.11 to 7.75] | 2.76 [1.45 to 6.87] | 11.99 [5.52 to 16.92] | 2.76 [2.07 to 2.79] | 6.90 [5.55 to 17.31] | 9.79 [5.75 to 16.36] | 6.60 [4.70 to 8.18] | 11.07 [6.87 to 15.18]

9. Secondary Outcome: Overall Survival (OS)
Description: Time from start of treatment to the date of death due to any cause. If the patient was alive at the date of the analysis cut-off or lost to follow-up, then OS was censored at the last contact date prior to data cut-off date.
  The Kaplan-Meier method was used to estimate OS, and the median OS, along with 95% confidence intervals, was reported.
Time Frame: Up to approximately 6 years
Population: FAS, including all subjects who received at least one dose of capmatinib.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1a: Pre-treated Patients With MET GCN ≥ 10 (2/3L) | Cohort 1b: Pre-treated Patients With MET GCN ≥ 6 and < 10 (2/3L) | Cohort 2: Pre-treated Patients With MET GCN ≥ 4 and < 6 (2/3L) | Cohort 3: Pre-treated Patients With MET GCN < 4 (2/3L) | Cohort 4: Pre-treated Patients With MET Mutation Regardless of MET GCN (2/3L) | Cohort 5a: Treatment-naïve Patients With MET GCN ≥10 (1L) | Cohort 5b: Treatment-naïve Patients With MET Mutation Regardless of MET GCN (1L) | Cohort 6.1 (Expansion of Cohort 1a): Pre-treated Patients MET GCN ≥ 10 Without MET Mutation (2L) | Cohort 6.2 (Expansion of Cohort 4): Pre-treated Patients With MET Mutation (2L) | Cohort 7 (Expansion of Cohort 5b): Treatment-naïve With MET Mutation Regardless of MET GCN (1L) | Cohort 4 + Cohort 6.2: All Pre-treated Patients With MET Mutation Regardless of MET GCN (2/3L) | Cohort 5b + Cohort 7: All Treatment-naive With MET Mutation Regardless of MET GCN (1L)
Number analyzed (Participants) | 69 | 42 | 54 | 30 | 69 | 15 | 28 | 3 | 31 | 32 | 100 | 60
Months | 10.61 [6.28 to 17.22] | 7.46 [5.59 to 10.18] | 10.15 [5.52 to 15.74] | 9.46 [4.11 to 12.32] | 13.57 [8.61 to 22.24] | 9.56 [4.80 to NA] — NA: not estimable due to the insufficient number of participants with events | 20.76 [12.42 to 43.93] | 4.14 [2.07 to NA] — NA: not estimable due to the insufficient number of participants with events | 25.95 [13.54 to 43.40] | 21.36 [12.85 to 34.76] | 16.79 [11.63 to 23.82] | 21.36 [15.24 to 30.52]

10. Secondary Outcome: Pharmacokinetic (PK) Concentrations of Capmatinib
Description: PK concentrations of capmatinib. Plasma concentrations of capmatinib were measured using validated liquid chromatography-tandem mass spectrometry (LCMS/MS) methods with a lower limit of quantification (LLOQ) of approximately 1.0 ng/mL.
  Capmatinib concentration data was summarized for Cohorts 1a, 1b, 2, 3, 4, 5a and 5b when capmatinib was administered in fasted state; and for Cohorts 6 and 7 when capmatinib was administered with or without food.
Time Frame: Cycle (C) 1 Day (D) 1 predose and 2 hours post-dose, C1D15 pre-dose and 2 hours post-dose, C3D1 pre-dose. Each Cycle is 21 days
Population: Participants who received at least one dose of capmatinib and provided at least one evaluable pharmacokinetic concentration for capmatinib at the specified time points. Participants who received capmatinib under the same administration conditions (fasted state or with/without food) were pooled together.
Measure: Mean (Standard Deviation); unit: nanogram/mililiter (ng/ml)
Groups:
- Cohorts 1-5: Capmatinib Administration in Fasted State: Participants from Cohorts 1a, 1b, 2, 3, 4, 5a and 5b who received capmatinib in fasted state
- Cohorts 6-7: Capmatinib Administration With ot Without Food: Participants from Cohorts 6 and 7 who received capmatinib with or without food
Arm/Group | Cohorts 1-5: Capmatinib Administration in Fasted State | Cohorts 6-7: Capmatinib Administration With ot Without Food
Number analyzed (Participants) | 275 | 54
nanogram/mililiter (ng/ml)
  Cycle 1 Day 1- pre-dose | 0.00 (0.00) | 0.00 (0.00)
  Cycle 1 Day 1- 2 hours post-dose: number analyzed (Participants) | 275 | 53
  Cycle 1 Day 1- 2 hours post-dose | 3360 (1920) | 3060 (1780)
  Cycle 1 Day 15 - pre-dose: number analyzed (Participants) | 176 | 29
  Cycle 1 Day 15 - pre-dose | 727 (781) | 663 (806)
  Cycle 1 Day 15- 2 hours post-dose: number analyzed (Participants) | 209 | 47
  Cycle 1 Day 15- 2 hours post-dose | 4100 (2100) | 4340 (2000)
  Cycle 3 Day 1 - pre-dose: number analyzed (Participants) | 96 | 18
  Cycle 3 Day 1 - pre-dose | 687 (1000) | 672 (745)

11. Secondary Outcome: Maximum Concentration (Cmax) of Capmatinib
Description: Cmax of capmatinib was estimated by non-compartmental analysis. Cmax is the maximum plasma drug concentration after single dose administration. Plasma concentrations of capmatinib were measured using validated LCMS/MS methods with a LLOQ of approximately 1.0 ng/mL.
  Only a subset of participants from Cohorts 1a, 1b, 2, 3, 4, 5a and 5b, who had an extensive PK collection schedule, were included in this analysis
Time Frame: Cycle 1 Day 1 and Day 15 at pre-dose, 0.5, 1, 2, 4, 6 and 8 hours post-dose. Each Cycle is 21 days
Population: Participants from Cohorts 1a, 1b, 2, 3, 4, 5a and 5b who received at least one dose of capmatinib with extensive PK sampling collection and an evaluable PK parameter (Cmax for capmatinib) at the specified time points. Participants received capmatinib under the same administration conditions (fasted state) and were pooled together for analysis
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Cohorts 1-5: Capmatinib Administration in Fasted State
Number analyzed (Participants) | 55
ng/ml
  Cycle 1 Day 1 | 4230 (2290)
  Cycle 1 Day 15: number analyzed (Participants) | 44
  Cycle 1 Day 15 | 5450 (2560)

12. Secondary Outcome: Maximum Concentration (Cmax) of CMN288
Description: Cmax of CMN288 (metabolite of capmatinib) was estimated by non-compartmental analysis. Cmax is the maximum plasma drug concentration after single dose administration. Plasma concentrations of metabolite CMN288 were measured using validated LCMS/MS methods with a LLOQ of approximately 1.0 ng/mL.
  Only a subset of participants from Cohorts 1a, 1b, 2, 3, 4, 5a and 5b, who had an extensive PK collection schedule, were included in this analysis
Time Frame: Cycle 1 Day 1 and Day 15 at pre-dose, 0.5, 1, 2, 4, 6 and 8 hours post-dose. Each Cycle is 21 days
Population: Participants from Cohorts 1a, 1b, 2, 3, 4, 5a and 5b who received at least one dose of capmatinib with extensive PK sampling collection and an evaluable PK parameter (Cmax for CMN288) at the specified time points. Participants received capmatinib under the same administration conditions (fasted state) and were pooled together for analysis
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Cohorts 1-5: Capmatinib Administration in Fasted State
Number analyzed (Participants) | 51
ng/ml
  Cycle 1 Day 1 | 1910 (1420)
  Cycle 1 Day 15: number analyzed (Participants) | 42
  Cycle 1 Day 15 | 1420 (725)

13. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Zero to Time Infinity (AUCinf) of Capmatinib
Description: AUCinf of capmatinib was estimated by non-compartmental analysis. AUCinf is the area under the plasma concentration-time curve extrapolated to infinity. Plasma concentrations of capmatinib were measured using validated LCMS/MS methods with a LLOQ of approximately 1.0 ng/mL.
  Only a subset of participants from Cohorts 1a, 1b, 2, 3, 4, 5a and 5b, who had an extensive PK collection schedule, were included in this analysis
Time Frame: Cycle 1 Day 1 at pre-dose, 0.5, 1, 2, 4, 6 and 8 hours post-dose. Each Cycle is 21 days
Population: Participants from Cohorts 1a, 1b, 2, 3, 4, 5a and 5b who received at least one dose of capmatinib with extensive PK sampling collection and an evaluable PK parameter (AUCinf for capmatinib) at the specified time points. Participants received capmatinib under the same administration conditions (fasted state) and were pooled together for analysis
Measure: Mean (Standard Deviation); unit: nanogram * hour / mililiter (ng*h/ml)
Arm/Group | Cohorts 1-5: Capmatinib Administration in Fasted State
Number analyzed (Participants) | 44
nanogram * hour / mililiter (ng*h/ml) | 17000 (7770)

14. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Zero to Time Infinity (AUCinf) of CMN288
Description: AUCinf of CMN288 (metabolite of capmatinib) was estimated by non-compartmental analysis. AUCinf is the area under the plasma concentration-time curve extrapolated to infinity. Plasma concentrations of metabolite CMN288 were measured using validated LCMS/MS methods with a LLOQ of approximately 1.0 ng/mL.
  Only a subset of participants from Cohorts 1a, 1b, 2, 3, 4, 5a and 5b, who had an extensive PK collection schedule, were included in this analysis
Time Frame: Cycle 1 Day 1 at pre-dose, 0.5, 1, 2, 4, 6 and 8 hours post-dose. Each Cycle is 21 days
Population: Participants from Cohorts 1a, 1b, 2, 3, 4, 5a and 5b who received at least one dose of capmatinib with extensive PK sampling collection and an evaluable PK parameter (AUCinf for CMN288) at the specified time points. Participants received capmatinib under the same administration conditions (fasted state) and were pooled together for analysis
Measure: Mean (Standard Deviation); unit: ng*h/ml
Arm/Group | Cohorts 1-5: Capmatinib Administration in Fasted State
Number analyzed (Participants) | 27
ng*h/ml | 9020 (5060)

15. Secondary Outcome: Time to Reach Maximum Concentration (Tmax) of Capmatinib
Description: Tmax of capmatinib was estimated by non-compartmental analysis. Tmax is the time to reach maximum plasma concentration. Actual recorded sampling times were considered for the calculations. Plasma concentrations of capmatinib were measured using validated LCMS/MS methods with a LLOQ of approximately 1.0 ng/mL.
  Only a subset of participants from Cohorts 1a, 1b, 2, 3, 4, 5a and 5b, who had an extensive PK collection schedule, were included in this analysis
Time Frame: Cycle 1 Day 1 and Day 15 at pre-dose, 0.5, 1, 2, 4, 6 and 8 hours post-dose. Each Cycle is 21 days
Population: Participants from Cohorts 1a, 1b, 2, 3, 4, 5a and 5b who received at least one dose of capmatinib with extensive PK sampling collection and an evaluable PK parameter (Tmax for capmatinib) at the specified time points. Participants received capmatinib under the same administration conditions (fasted state) and were pooled together for analysis
Measure: Median (Full Range); unit: hour
Arm/Group | Cohorts 1-5: Capmatinib Administration in Fasted State
Number analyzed (Participants) | 55
hour
  Cycle 1 Day 1 | 1.87 [0.583 to 4.03]
  Cycle 1 Day 15: number analyzed (Participants) | 44
  Cycle 1 Day 15 | 1.09 [0.5 to 6.07]

16. Secondary Outcome: Time to Reach Maximum Concentration (Tmax) of CMN288
Description: Tmax of CMN288 (metabolite of capmatinib) was estimated by non-compartmental analysis. Tmax is the time to reach maximum plasma concentration. Actual recorded sampling times were considered for the calculations. Plasma concentrations of metabolite CMN288 were measured using validated LCMS/MS methods with a LLOQ of approximately 1.0 ng/mL.
  Only a subset of participants from cohorts 1-5, who had an extensive PK collection schedule, were included in this analysis
Time Frame: Cycle 1 Day 1 and Day 15 at pre-dose, 0.5, 1, 2, 4, 6 and 8 hours post-dose. Each Cycle is 21 days
Population: Participants from Cohorts 1a, 1b, 2, 3, 4, 5a and 5b who received at least one dose of capmatinib with extensive PK sampling collection and an evaluable PK parameter (Tmax for CMN288) at the specified time points. Participants received capmatinib under the same administration conditions (fasted state) and were pooled together for analysis
Measure: Median (Full Range); unit: hour
Arm/Group | Cohorts 1-5: Capmatinib Administration in Fasted State
Number analyzed (Participants) | 51
hour
  Cycle 1 Day 1 | 1.93 [0.950 to 4.03]
  Cycle 1 Day 15: number analyzed (Participants) | 42
  Cycle 1 Day 15 | 1.91 [0.883 to 7.98]

17. Secondary Outcome: Elimination Half-life (T1/2) of Capmatinib
Description: T1/2 of capmatinib was estimated by non-compartmental analysis. T1/2 is the time it takes for the concentration of capmatinib in the bloodstream to decrease by half. Plasma concentrations of capmatinib were measured using validated LCMS/MS methods with a LLOQ of approximately 1.0 ng/mL.
  Only a subset of participants from Cohorts 1a, 1b, 2, 3, 4, 5a and 5b, who had an extensive PK collection schedule, were included in this analysis
Time Frame: Cycle 1 Day 1 and Day 15 at pre-dose, 0.5, 1, 2, 4, 6 and 8 hours post-dose. Each Cycle is 21 days
Population: Participants from Cohorts 1a, 1b, 2, 3, 4, 5a and 5b who received at least one dose of capmatinib with extensive PK sampling collection and an evaluable PK parameter (T1/2 for capmatinib) at the specified time points. Participants received capmatinib under the same administration conditions (fasted state) and were pooled together for analysis
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Cohorts 1-5: Capmatinib Administration in Fasted State
Number analyzed (Participants) | 47
hour
  Cycle 1 Day 1 | 1.87 (0.947)
  Cycle 1 Day 15: number analyzed (Participants) | 37
  Cycle 1 Day 15 | 2.40 (0.652)

18. Secondary Outcome: Elimination Half-life (T1/2) of CMN288
Description: T1/2 of CMN288 (metabolite of capmatinib) was estimated by non-compartmental analysis. T1/2 is the time it takes for the concentration of CMN288 in the bloodstream to decrease by half. Plasma concentrations of metabolite CMN288 were measured using validated LCMS/MS methods with a LLOQ of approximately 1.0 ng/mL.
  Only a subset of participants from Cohorts 1a, 1b, 2, 3, 4, 5a and 5b, who had an extensive PK collection schedule, were included in this analysis
Time Frame: Cycle 1 Day 1 and Day 15 at pre-dose, 0.5, 1, 2, 4, 6 and 8 hours post-dose. Each Cycle is 21 days
Population: Participants from Cohorts 1a, 1b, 2, 3, 4, 5a and 5b who received at least one dose of capmatinib with extensive PK sampling collection and an evaluable PK parameter (T1/2 for CMN288) at the specified time points. Participants received capmatinib under the same administration conditions (fasted state) and were pooled together for analysis
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Cohorts 1-5: Capmatinib Administration in Fasted State
Number analyzed (Participants) | 40
hour
  Cycle 1 Day 1 | 3.14 (1.42)
  Cycle 1 Day 15: number analyzed (Participants) | 34
  Cycle 1 Day 15 | 3.06 (0.949)

19. Post Hoc Outcome: All Collected Deaths
Description: On-treatment deaths were collected from start of treatment to 30 days after last dose of treatment.
  Post-treatment efficacy/survival follow-up deaths were collected from 31 days after last dose of treatment until the end of the study.
  All deaths refer to the sum of on-treatment and post-treatment efficacy/survival follow-up deaths.
Time Frame: On-treatment: Up to approximately 5.5 years. Post-treatment efficacy/survival follow-up: Up to approximately 6 years
Population: FAS, including all subjects who received at least one dose of capmatinib
Measure: Number; unit: Participants
Groups:
- All Participants: All participants
Arm/Group | Cohort 1a: Pre-treated Patients With MET GCN ≥ 10 (2/3L) | Cohort 1b: Pre-treated Patients With MET GCN ≥ 6 and < 10 (2/3L) | Cohort 2: Pre-treated Patients With MET GCN ≥ 4 and < 6 (2/3L) | Cohort 3: Pre-treated Patients With MET GCN < 4 (2/3L) | Cohort 4: Pre-treated Patients With MET Mutation Regardless of MET GCN (2/3L) | Cohort 5a: Treatment-naïve Patients With MET GCN ≥10 (1L) | Cohort 5b: Treatment-naïve Patients With MET Mutation Regardless of MET GCN (1L) | Cohort 6.1 (Expansion of Cohort 1a): Pre-treated Patients MET GCN ≥ 10 Without MET Mutation (2L) | Cohort 6.2 (Expansion of Cohort 4): Pre-treated Patients With MET Mutation (2L) | Cohort 7 (Expansion of Cohort 5b): Treatment-naïve With MET Mutation Regardless of MET GCN (1L) | Cohort 4 + Cohort 6.2: All Pre-treated Patients With MET Mutation Regardless of MET GCN (2/3L) | Cohort 5b + Cohort 7: All Treatment-naive With MET Mutation Regardless of MET GCN (1L) | All Participants
Number analyzed (Participants) | 69 | 42 | 54 | 30 | 69 | 15 | 28 | 3 | 31 | 32 | 100 | 60 | 373
Participants
  On-treatment | 10 | 7 | 12 | 4 | 14 | 0 | 5 | 1 | 5 | 5 | 19 | 10 | 63
  Post-treatment efficacy/survival follow-up: number analyzed (Participants) | 59 | 35 | 42 | 25 | 55 | 15 | 20 | 2 | 20 | 23 | 75 | 43 | 296
  Post-treatment efficacy/survival follow-up | 44 | 26 | 34 | 22 | 44 | 13 | 13 | 2 | 17 | 16 | 61 | 29 | 231
  All deaths | 54 | 33 | 46 | 26 | 58 | 13 | 18 | 3 | 22 | 21 | 80 | 39 | 294

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from first dose of study treatment to 30 days after last dose of study medication (on-treatment), up to approximately 5.5 years. Deaths were collected in the post treatment efficacy/survival follow-up from 31 days after last dose of study medication until the end of the study, up to approximately 6 years.
Description: Deaths in the post-treatment efficacy/survival follow-up are not counted as AEs. The total number at risk in the post-treatment efficacy/survival includes patients who entered the post-treatment efficacy and/or survival follow-up periods.
Groups:
- Cohort 1a: On-treatment; Cohort 1b: On-treatment; All Patients: On-treatment: AEs collected during the on-treatment period (up to 30 days post-treatment)
- Cohort 2: On-treatment; Cohort 3: On-treatment; Cohort 4: On-treatment; Cohort 5a: On-treatment; Cohort 5b: On-treatment; Cohort 6.1 (Expansion of Cohort 1a): On-treatment; Cohort 6.2 (Expansion of Cohort 4): On-treatment; Cohort 7 (Expansion of Cohort 5b): On-treatment; Cohort 4 + Cohort 6.2: On-treatment; Cohort 5b + Cohort 7: On-treatment: AEs collected during on-treatment period (up to 30 days post-treatment)
- Cohort 1a: Post-treatment Efficacy/Survival Follow-up; Cohort 1b: Post-treatment Efficacy/Survival Follow-up Period; All Patients: Post-treatment Efficacy/Survival Follow-up: Deaths collected in the post- treatment efficacy/survival follow-up period (starting from day 31 post- treatment). No AEs were collected during this period
- Cohort 2: Post-treatment Efficacy/Survival Follow-up Period; Cohort 3: Post-treatment Efficacy/Survival Follow-up Period; Cohort 4: Post-treatment Efficacy/Survival Follow-up Period; Cohort 5a: Post-treatment Efficacy/Survival Follow-up Period; Cohort 5b: Post-treatment Efficacy/Survival Follow-up Period; Cohort 6.1 (Expansion of Cohort 1a): Post-treatment Efficacy/Survival Follow-up Period; Cohort 6.2 (Expansion of Cohort 4): Post-treatment Efficacy/Survival Follow-up Period; Cohort 7 (Expansion of Cohort 5b): Post-treatment Efficacy/Survival Follow-up Period; Cohort 4 + Cohort 6.2: Post-treatment Efficacy/Survival Follow-up Period; Cohort 5b + Cohort 7: Post-treatment Efficacy/Survival Follow-up Period: Deaths collected in the post-treatment efficacy/survival follow-up period (starting from day 31 post- treatment). No AEs were collected during this period
Arm/Group | Cohort 1a: On-treatment | Cohort 1b: On-treatment | Cohort 2: On-treatment | Cohort 3: On-treatment | Cohort 4: On-treatment | Cohort 5a: On-treatment | Cohort 5b: On-treatment | Cohort 6.1 (Expansion of Cohort 1a): On-treatment | Cohort 6.2 (Expansion of Cohort 4): On-treatment | Cohort 7 (Expansion of Cohort 5b): On-treatment | Cohort 4 + Cohort 6.2: On-treatment | Cohort 5b + Cohort 7: On-treatment | All Patients: On-treatment | Cohort 1a: Post-treatment Efficacy/Survival Follow-up | Cohort 1b: Post-treatment Efficacy/Survival Follow-up Period | Cohort 2: Post-treatment Efficacy/Survival Follow-up Period | Cohort 3: Post-treatment Efficacy/Survival Follow-up Period | Cohort 4: Post-treatment Efficacy/Survival Follow-up Period | Cohort 5a: Post-treatment Efficacy/Survival Follow-up Period | Cohort 5b: Post-treatment Efficacy/Survival Follow-up Period | Cohort 6.1 (Expansion of Cohort 1a): Post-treatment Efficacy/Survival Follow-up Period | Cohort 6.2 (Expansion of Cohort 4): Post-treatment Efficacy/Survival Follow-up Period | Cohort 7 (Expansion of Cohort 5b): Post-treatment Efficacy/Survival Follow-up Period | Cohort 4 + Cohort 6.2: Post-treatment Efficacy/Survival Follow-up Period | Cohort 5b + Cohort 7: Post-treatment Efficacy/Survival Follow-up Period | All Patients: Post-treatment Efficacy/Survival Follow-up
All-Cause Mortality (participants affected / at risk) | 10/69 | 7/42 | 12/54 | 4/30 | 14/69 | 0/15 | 5/28 | 1/3 | 5/31 | 5/32 | 19/100 | 10/60 | 63/373 | 44/59 | 26/35 | 34/42 | 22/25 | 44/55 | 13/15 | 13/20 | 2/2 | 17/20 | 16/23 | 61/75 | 29/43 | 231/296
Serious Adverse Events (participants affected / at risk) | 42/69 | 21/42 | 30/54 | 15/30 | 38/69 | 9/15 | 14/28 | 2/3 | 14/31 | 17/32 | 52/100 | 31/60 | 202/373 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 66/69 | 41/42 | 53/54 | 28/30 | 66/69 | 15/15 | 28/28 | 3/3 | 29/31 | 31/32 | 95/100 | 59/60 | 360/373 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1a: On-treatment (N=69) | Cohort 1b: On-treatment (N=42) | Cohort 2: On-treatment (N=54) | Cohort 3: On-treatment (N=30) | Cohort 4: On-treatment (N=69) | Cohort 5a: On-treatment (N=15) | Cohort 5b: On-treatment (N=28) | Cohort 6.1 (Expansion of Cohort 1a): On-treatment (N=3) | Cohort 6.2 (Expansion of Cohort 4): On-treatment (N=31) | Cohort 7 (Expansion of Cohort 5b): On-treatment (N=32) | Cohort 4 + Cohort 6.2: On-treatment (N=100) | Cohort 5b + Cohort 7: On-treatment (N=60) | All Patients: On-treatment (N=373) | Cohort 1a: Post-treatment Efficacy/Survival Follow-up (N=0) | Cohort 1b: Post-treatment Efficacy/Survival Follow-up Period (N=0) | Cohort 2: Post-treatment Efficacy/Survival Follow-up Period (N=0) | Cohort 3: Post-treatment Efficacy/Survival Follow-up Period (N=0) | Cohort 4: Post-treatment Efficacy/Survival Follow-up Period (N=0) | Cohort 5a: Post-treatment Efficacy/Survival Follow-up Period (N=0) | Cohort 5b: Post-treatment Efficacy/Survival Follow-up Period (N=0) | Cohort 6.1 (Expansion of Cohort 1a): Post-treatment Efficacy/Survival Follow-up Period (N=0) | Cohort 6.2 (Expansion of Cohort 4): Post-treatment Efficacy/Survival Follow-up Period (N=0) | Cohort 7 (Expansion of Cohort 5b): Post-treatment Efficacy/Survival Follow-up Period (N=0) | Cohort 4 + Cohort 6.2: Post-treatment Efficacy/Survival Follow-up Period (N=0) | Cohort 5b + Cohort 7: Post-treatment Efficacy/Survival Follow-up Period (N=0) | All Patients: Post-treatment Efficacy/Survival Follow-up (N=0)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 2 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Cardiac failure (Cardiac disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 4 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Cardiopulmonary failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Spinal muscular atrophy (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 2 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Primary adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 6 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Anal prolapse (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 3 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Duodenal stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Duodenitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Dysphagia (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Intestinal polyp (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Nausea (Gastrointestinal disorders) | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 7 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Oesophageal stenosis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Vomiting (Gastrointestinal disorders) | 4 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 9 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Asthenia (General disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Drug withdrawal syndrome (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
General physical health deterioration (General disorders) | 3 | 3 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 11 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Generalised oedema (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Malaise (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Non-cardiac chest pain (General disorders) | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 4 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Oedema peripheral (General disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 3 | 6 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Peripheral swelling (General disorders) | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 4 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pyrexia (General disorders) | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 5 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Stenosis (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Vascular device occlusion (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 2 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hepatitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 4 | 0 | 1 | 0 | 0 | 0 | 4 | 1 | 6 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Device related infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 2 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Haemophilus infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Infectious pleural effusion (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Influenza (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Lung abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Medical device site infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pleural infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pneumonia (Infections and infestations) | 7 | 4 | 3 | 1 | 4 | 0 | 0 | 1 | 2 | 1 | 6 | 1 | 23 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pneumonia aspiration (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pneumonia influenzal (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Respiratory tract infection (Infections and infestations) | 1 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Accidental exposure to product (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 3 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Fracture displacement (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Radiation necrosis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Amylase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Eastern Cooperative Oncology Group performance status worsened (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
General physical condition abnormal (Investigations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Troponin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 1 | 3 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 2 | 6 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 4 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 3 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Osteolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 3 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Aphasia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Cerebral ischaemia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Cerebral mass effect (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Epilepsy (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hemiparesis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Neurological symptom (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Paraplegia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Seizure (Nervous system disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Disorientation (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Organic brain syndrome (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Calculus urinary (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Renal failure (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Renal infarct (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Breast pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Genital prolapse (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Scrotal oedema (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 4 | 3 | 2 | 6 | 1 | 2 | 0 | 1 | 1 | 7 | 3 | 26 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 2 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 | 1 | 3 | 0 | 2 | 1 | 0 | 0 | 1 | 2 | 3 | 2 | 16 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 1 | 3 | 2 | 6 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 4 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 7 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pulmonary venous thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 5 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Embolism (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Jugular vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Peripheral ischaemia (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Superior vena cava syndrome (Vascular disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Venous thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1a: On-treatment (N=69) | Cohort 1b: On-treatment (N=42) | Cohort 2: On-treatment (N=54) | Cohort 3: On-treatment (N=30) | Cohort 4: On-treatment (N=69) | Cohort 5a: On-treatment (N=15) | Cohort 5b: On-treatment (N=28) | Cohort 6.1 (Expansion of Cohort 1a): On-treatment (N=3) | Cohort 6.2 (Expansion of Cohort 4): On-treatment (N=31) | Cohort 7 (Expansion of Cohort 5b): On-treatment (N=32) | Cohort 4 + Cohort 6.2: On-treatment (N=100) | Cohort 5b + Cohort 7: On-treatment (N=60) | All Patients: On-treatment (N=373) | Cohort 1a: Post-treatment Efficacy/Survival Follow-up (N=0) | Cohort 1b: Post-treatment Efficacy/Survival Follow-up Period (N=0) | Cohort 2: Post-treatment Efficacy/Survival Follow-up Period (N=0) | Cohort 3: Post-treatment Efficacy/Survival Follow-up Period (N=0) | Cohort 4: Post-treatment Efficacy/Survival Follow-up Period (N=0) | Cohort 5a: Post-treatment Efficacy/Survival Follow-up Period (N=0) | Cohort 5b: Post-treatment Efficacy/Survival Follow-up Period (N=0) | Cohort 6.1 (Expansion of Cohort 1a): Post-treatment Efficacy/Survival Follow-up Period (N=0) | Cohort 6.2 (Expansion of Cohort 4): Post-treatment Efficacy/Survival Follow-up Period (N=0) | Cohort 7 (Expansion of Cohort 5b): Post-treatment Efficacy/Survival Follow-up Period (N=0) | Cohort 4 + Cohort 6.2: Post-treatment Efficacy/Survival Follow-up Period (N=0) | Cohort 5b + Cohort 7: Post-treatment Efficacy/Survival Follow-up Period (N=0) | All Patients: Post-treatment Efficacy/Survival Follow-up (N=0)
Anaemia (Blood and lymphatic system disorders) | 5 | 2 | 5 | 6 | 8 | 1 | 2 | 0 | 4 | 2 | 12 | 4 | 35 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 6 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 5 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 1 | 1 | 1 | 1 | 2 | 0 | 1 | 0 | 2 | 2 | 9 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 3 | 3 | 5 | 3 | 9 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Atrial fibrillation (Cardiac disorders) | 2 | 0 | 2 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 2 | 1 | 8 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Cardiac failure (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 3 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Palpitations (Cardiac disorders) | 1 | 1 | 1 | 0 | 2 | 1 | 1 | 0 | 0 | 2 | 2 | 3 | 9 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 4 | 0 | 1 | 0 | 0 | 0 | 4 | 1 | 5 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Tachycardia (Cardiac disorders) | 0 | 3 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 5 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hypoacusis (Ear and labyrinth disorders) | 2 | 1 | 1 | 0 | 3 | 0 | 2 | 0 | 0 | 5 | 3 | 7 | 14 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 3 | 1 | 3 | 4 | 8 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Vertigo (Ear and labyrinth disorders) | 2 | 2 | 2 | 2 | 5 | 0 | 1 | 0 | 1 | 0 | 6 | 1 | 15 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hyperthyroidism (Endocrine disorders) | 1 | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 7 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 5 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Abdominal pain (Gastrointestinal disorders) | 2 | 3 | 7 | 1 | 3 | 0 | 3 | 0 | 1 | 3 | 4 | 6 | 23 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Abdominal pain upper (Gastrointestinal disorders) | 4 | 4 | 2 | 2 | 5 | 0 | 5 | 0 | 2 | 3 | 7 | 8 | 27 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Abnormal faeces (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Constipation (Gastrointestinal disorders) | 16 | 9 | 10 | 7 | 9 | 6 | 5 | 1 | 3 | 3 | 12 | 8 | 69 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Diarrhoea (Gastrointestinal disorders) | 18 | 6 | 7 | 8 | 13 | 4 | 5 | 0 | 5 | 4 | 18 | 9 | 70 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 5 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Dyspepsia (Gastrointestinal disorders) | 4 | 3 | 4 | 3 | 6 | 0 | 2 | 1 | 1 | 2 | 7 | 4 | 26 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Dysphagia (Gastrointestinal disorders) | 2 | 4 | 6 | 1 | 1 | 2 | 0 | 0 | 0 | 1 | 1 | 1 | 17 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 1 | 3 | 0 | 1 | 0 | 1 | 0 | 1 | 2 | 2 | 3 | 12 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Nausea (Gastrointestinal disorders) | 32 | 16 | 24 | 15 | 32 | 9 | 13 | 2 | 12 | 15 | 44 | 28 | 170 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 3 | 0 | 3 | 1 | 0 | 0 | 1 | 2 | 4 | 2 | 11 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Vomiting (Gastrointestinal disorders) | 22 | 14 | 12 | 9 | 19 | 4 | 7 | 1 | 8 | 6 | 27 | 13 | 102 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Asthenia (General disorders) | 6 | 8 | 11 | 3 | 6 | 2 | 4 | 0 | 3 | 6 | 9 | 10 | 49 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Chest discomfort (General disorders) | 1 | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 6 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Face oedema (General disorders) | 1 | 0 | 1 | 0 | 4 | 0 | 2 | 0 | 1 | 0 | 5 | 2 | 9 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Fatigue (General disorders) | 11 | 10 | 16 | 6 | 19 | 2 | 4 | 1 | 11 | 6 | 30 | 10 | 86 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Generalised oedema (General disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 2 | 2 | 3 | 6 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Malaise (General disorders) | 2 | 0 | 1 | 0 | 3 | 0 | 2 | 0 | 1 | 0 | 4 | 2 | 9 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Non-cardiac chest pain (General disorders) | 8 | 5 | 7 | 1 | 4 | 3 | 1 | 0 | 3 | 0 | 7 | 1 | 32 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Oedema (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 3 | 0 | 7 | 8 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Oedema peripheral (General disorders) | 34 | 18 | 24 | 11 | 38 | 10 | 21 | 1 | 23 | 23 | 61 | 44 | 203 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pain (General disorders) | 4 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 9 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Peripheral swelling (General disorders) | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 3 | 1 | 4 | 10 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pyrexia (General disorders) | 8 | 7 | 8 | 5 | 9 | 3 | 2 | 1 | 2 | 4 | 11 | 6 | 49 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hepatic steatosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Contrast media allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 3 | 3 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Bronchitis (Infections and infestations) | 1 | 1 | 3 | 0 | 4 | 0 | 0 | 0 | 1 | 0 | 5 | 0 | 10 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 3 | 3 | 4 | 7 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Cellulitis (Infections and infestations) | 3 | 0 | 1 | 0 | 4 | 0 | 2 | 0 | 3 | 0 | 7 | 2 | 13 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Epididymitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 2 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Erysipelas (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 2 | 4 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 2 | 1 | 4 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Influenza (Infections and infestations) | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 5 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Nasopharyngitis (Infections and infestations) | 7 | 4 | 1 | 1 | 3 | 1 | 2 | 0 | 3 | 2 | 6 | 4 | 24 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Oral candidiasis (Infections and infestations) | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 5 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pneumonia (Infections and infestations) | 6 | 5 | 1 | 3 | 5 | 1 | 2 | 0 | 2 | 2 | 7 | 4 | 27 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pyuria (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 2 | 5 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Urinary tract infection (Infections and infestations) | 0 | 1 | 1 | 0 | 7 | 0 | 0 | 0 | 2 | 2 | 9 | 2 | 13 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Anastomotic ulcer (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Face injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 2 | 1 | 2 | 0 | 2 | 2 | 4 | 4 | 11 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 3 | 1 | 4 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Alanine aminotransferase increased (Investigations) | 13 | 4 | 5 | 3 | 9 | 5 | 4 | 0 | 7 | 3 | 16 | 7 | 53 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Amylase increased (Investigations) | 9 | 3 | 2 | 1 | 7 | 3 | 2 | 0 | 4 | 5 | 11 | 7 | 36 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Aspartate aminotransferase increased (Investigations) | 11 | 2 | 4 | 3 | 6 | 5 | 2 | 0 | 4 | 2 | 10 | 4 | 39 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Blood albumin decreased (Investigations) | 3 | 0 | 1 | 1 | 5 | 1 | 0 | 0 | 0 | 2 | 5 | 2 | 13 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Blood alkaline phosphatase increased (Investigations) | 8 | 1 | 3 | 0 | 5 | 1 | 1 | 0 | 3 | 3 | 8 | 4 | 25 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Blood bilirubin increased (Investigations) | 3 | 2 | 1 | 1 | 1 | 0 | 2 | 0 | 1 | 2 | 2 | 4 | 13 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Blood creatinine increased (Investigations) | 16 | 8 | 14 | 5 | 24 | 3 | 10 | 1 | 10 | 12 | 34 | 22 | 103 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Blood urine present (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
C-reactive protein increased (Investigations) | 3 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 2 | 9 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Eastern Cooperative Oncology Group performance status worsened (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Gamma-glutamyltransferase increased (Investigations) | 9 | 2 | 5 | 0 | 3 | 0 | 2 | 0 | 3 | 0 | 6 | 2 | 24 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Lipase increased (Investigations) | 5 | 4 | 1 | 4 | 7 | 1 | 5 | 0 | 3 | 7 | 10 | 12 | 37 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Liver function test increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 1 | 2 | 4 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Lymphocyte count decreased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 1 | 3 | 5 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Neutrophil count decreased (Investigations) | 3 | 0 | 2 | 1 | 2 | 1 | 1 | 0 | 1 | 3 | 3 | 4 | 14 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Platelet count decreased (Investigations) | 3 | 0 | 3 | 1 | 5 | 1 | 1 | 1 | 1 | 1 | 6 | 2 | 17 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Procalcitonin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Protein total decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 1 | 3 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Weight decreased (Investigations) | 7 | 4 | 2 | 4 | 9 | 3 | 4 | 1 | 1 | 6 | 10 | 10 | 41 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Weight increased (Investigations) | 7 | 0 | 2 | 0 | 4 | 1 | 3 | 0 | 2 | 2 | 6 | 5 | 21 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
White blood cell count decreased (Investigations) | 2 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 1 | 1 | 2 | 8 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Decreased appetite (Metabolism and nutrition disorders) | 15 | 6 | 12 | 8 | 15 | 4 | 8 | 0 | 6 | 6 | 21 | 14 | 80 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 6 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1 | 4 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 9 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hypoalbuminaemia (Metabolism and nutrition disorders) | 9 | 4 | 5 | 0 | 5 | 1 | 3 | 0 | 6 | 5 | 11 | 8 | 38 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 5 | 1 | 3 | 0 | 4 | 8 | 9 | 11 | 23 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 2 | 2 | 3 | 3 | 1 | 1 | 0 | 2 | 4 | 5 | 5 | 23 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 2 | 2 | 7 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 2 | 3 | 0 | 3 | 2 | 1 | 1 | 0 | 2 | 3 | 3 | 15 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hypophagia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hypophosphataemia (Metabolism and nutrition disorders) | 9 | 0 | 1 | 0 | 3 | 0 | 3 | 0 | 4 | 0 | 7 | 3 | 20 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 3 | 7 | 0 | 8 | 3 | 7 | 1 | 2 | 2 | 10 | 9 | 39 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 7 | 10 | 2 | 11 | 2 | 4 | 1 | 11 | 7 | 22 | 11 | 63 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 2 | 1 | 5 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 1 | 2 | 6 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 6 | 3 | 1 | 1 | 3 | 3 | 0 | 2 | 3 | 3 | 6 | 26 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 3 | 2 | 4 | 3 | 10 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3 | 2 | 6 | 1 | 1 | 0 | 1 | 1 | 7 | 2 | 18 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 1 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 1 | 2 | 9 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 3 | 1 | 1 | 5 | 2 | 1 | 0 | 2 | 0 | 7 | 1 | 19 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 4 | 0 | 1 | 0 | 1 | 1 | 5 | 2 | 8 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 2 | 3 | 1 | 7 | 1 | 3 | 0 | 5 | 3 | 12 | 6 | 31 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Dizziness (Nervous system disorders) | 4 | 5 | 1 | 2 | 9 | 2 | 3 | 1 | 3 | 4 | 12 | 7 | 34 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Dysgeusia (Nervous system disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 3 | 6 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Headache (Nervous system disorders) | 6 | 4 | 3 | 2 | 9 | 1 | 2 | 0 | 2 | 1 | 11 | 3 | 30 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hypoaesthesia (Nervous system disorders) | 1 | 1 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 6 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 3 | 2 | 3 | 6 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Paraesthesia (Nervous system disorders) | 1 | 3 | 2 | 0 | 3 | 0 | 1 | 0 | 3 | 2 | 6 | 3 | 15 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Somnolence (Nervous system disorders) | 2 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 5 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Syncope (Nervous system disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 2 | 5 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Taste disorder (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 2 | 1 | 5 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Tremor (Nervous system disorders) | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 6 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Anxiety (Psychiatric disorders) | 0 | 3 | 4 | 0 | 3 | 1 | 2 | 0 | 1 | 1 | 4 | 3 | 15 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Confusional state (Psychiatric disorders) | 2 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 5 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Depression (Psychiatric disorders) | 1 | 1 | 2 | 0 | 3 | 0 | 0 | 0 | 3 | 2 | 6 | 2 | 12 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Dysphoria (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Insomnia (Psychiatric disorders) | 7 | 3 | 3 | 1 | 6 | 0 | 5 | 0 | 3 | 6 | 9 | 11 | 34 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Sleep disorder (Psychiatric disorders) | 1 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Dysuria (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 4 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Renal failure (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 2 | 3 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Breast swelling (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Oedema genital (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 3 | 3 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 9 | 9 | 4 | 11 | 2 | 7 | 0 | 7 | 3 | 18 | 10 | 61 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 0 | 1 | 2 | 0 | 1 | 0 | 2 | 0 | 4 | 1 | 11 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 | 15 | 11 | 5 | 16 | 5 | 6 | 2 | 6 | 6 | 22 | 12 | 83 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 3 | 1 | 1 | 0 | 0 | 1 | 3 | 2 | 8 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 3 | 2 | 1 | 0 | 0 | 3 | 3 | 4 | 11 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 3 | 0 | 1 | 0 | 1 | 1 | 3 | 1 | 4 | 2 | 16 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 2 | 0 | 4 | 1 | 5 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 3 | 0 | 4 | 0 | 8 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 3 | 0 | 3 | 0 | 0 | 0 | 2 | 2 | 5 | 2 | 17 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 2 | 2 | 3 | 5 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 1 | 4 | 0 | 1 | 1 | 0 | 1 | 4 | 2 | 11 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 2 | 4 | 4 | 0 | 3 | 0 | 1 | 2 | 5 | 5 | 19 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 2 | 0 | 2 | 2 | 2 | 0 | 0 | 2 | 2 | 4 | 15 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 1 | 3 | 2 | 5 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 2 | 0 | 1 | 0 | 2 | 1 | 4 | 2 | 9 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 3 | 2 | 4 | 10 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 2 | 3 | 2 | 7 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Dry skin (Skin and subcutaneous tissue disorders) | 9 | 1 | 2 | 1 | 2 | 2 | 0 | 0 | 1 | 1 | 3 | 1 | 19 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 3 | 1 | 4 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 6 | 3 | 0 | 10 | 2 | 2 | 0 | 3 | 2 | 13 | 4 | 35 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pruritus allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Rash (Skin and subcutaneous tissue disorders) | 3 | 1 | 4 | 1 | 6 | 2 | 0 | 0 | 4 | 3 | 10 | 3 | 24 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 6 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Skin induration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 4 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Deep vein thrombosis (Vascular disorders) | 0 | 2 | 2 | 0 | 1 | 1 | 0 | 0 | 1 | 2 | 2 | 2 | 9 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Embolism (Vascular disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 2 | 1 | 5 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hypertension (Vascular disorders) | 4 | 0 | 1 | 1 | 2 | 1 | 1 | 0 | 2 | 1 | 4 | 2 | 13 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hypotension (Vascular disorders) | 4 | 1 | 2 | 1 | 5 | 0 | 0 | 0 | 1 | 5 | 6 | 5 | 19 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Superficial vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 2 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-02-28): https://cdn.clinicaltrials.gov/large-docs/39/NCT02414139/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-03): https://cdn.clinicaltrials.gov/large-docs/39/NCT02414139/SAP_001.pdf